CLINICAL TRIAL: NCT03436888
Title: Cross-cultural Adaptation and Validation of the Pelvic Girdle Questionnaire in French Language
Acronym: PELVIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A00949-44
Record Dates: First submitted 2017-11-16; First posted 2018-02-19 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2022-02

CONDITIONS: Pelvic Girdle Pain; Pregnancy Related; Postpartum Period
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is the adaptation of the Pelvic Girdle Questionnaire to the French language from France, and the analysis of its psychometric properties. Firstly, a translation and adaptation process will be performed according to international guidelines. Secondly, the validation process will be performed through a sample of 250 pregnant or postpartum women suffering from pelvic girdle pain. They will fill several questionnaires, including Pelvic Girdle Questionnaire, that will allow us to analyse psychometric properties of the French version.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 years-old, pregnant or having given birth less than one year earlier, with PGP whose onset occurred during pregnancy or within 3 weeks after birth. Registered in the French social security system.

Exclusion Criteria:

* Ovarian cysts, uterine fibroids, caesarean section (if subject in postpartum period), radicular pain below the knee, previous surgery on the spine, pelvis or lower limbs, vaginismus-type pelvic pain, spondylolisthesis, inflammatory diseases, prolapse, suspected serious pathology (weakness of the lower limbs, reflex changes or loss of sensation associated with the same spinal nerve), impossibility or difficulty in understanding the questionnaires and subjects needing guardianship/supervision.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult pregnant or in postpartum period females suffering of pelvic girdle pain. The symptoms must occur during pregnancy or within 3 weeks after childbirth.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Disability | up to ten days
  Disability will be measured using Pelvic Girdle Questionnaire

SECONDARY OUTCOMES:
Disability: Oswestry disability index | 1 day (First appointment)
  Disability will be measured using Oswestry disability index
fear-avoidance beliefs: Fear Avoidance Beliefs Questionnaire | 1 day (First appointment)
  Fear Avoidance Beliefs will be measured using Fear Avoidance Beliefs Questionnaire
Pain Catastrophizing: Pain catastrophizing scale | 1 day (First appointment)
  Pain catastrophizing will be measured using pain catastrophizing scale
health-related quality of life: SF 8 scale | 1 day (First appointment)
  Health-related quality of life will be measured using SF 8 scale
Pain: Visual Analogue Pain Rating Scale | 1 day (First appointment)
  Pain will be measured using Visual Analogue Pain Rating Scale

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pôle de Santé de la Grâce de Dieu, Caen
  - Caen University Hospital, Caen

IPD SHARING:
Plan to Share IPD: No